CLINICAL TRIAL: NCT06056414
Title: Study of the Reduction of Anxiety After a Session of Energy Resonance by Cutaneous Stimulation in the Management of Patients Requiring Breast Macrobiopsy.
Brief Title: Study of Anxiety After a Session of Energy Resonance by Cutaneous Stimulation
Acronym: MBRESC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHB23.02
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Breast Neoplasm
Keywords: macrobiopsy; anxiety; Energy Resonance by Cutaneous Stimulation
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Energy Resonance by Cutaneous Stimulation (Experimental): one Energy Resonance by Cutaneous Stimulation session performed before macrobiopsy
  Interventions: Other: Energy Resonance by Cutaneous Stimulation

INTERVENTIONS:
Other: Energy Resonance by Cutaneous Stimulation — Energy Resonance by Cutaneous Stimulation session

SUMMARY:
Performing a breast macrobiopsy can be extremely delicate and anxiety-provoking. It can have an impact on the course of future examinations.

Patients' emotional feelings also have a definite impact on the nursing staff. The purpose of the MBRESC study is to evaluate Energy Resonance by Cutaneous Stimulation , a manual acupressure technique, in the management of anxiety prior to breast macrobiopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patient has received full information on the organization and purpose of the research, and has signed an informed consent form.
* Patient over 18 years of age
* Patient undergoing a diagnostic breast macrobiopsy for suspected breast cancer
* Patient undergoing a macro breast biopsy for the first time
* Patient affiliated to or benefiting from a social security schem

Exclusion Criteria:

* Patient with a history of breast cancer or other pathologies requiring invasive procedures
* Patient with several lesions to be biopsied
* Patient with psychiatric pathology
* Patient under anxiolytic or psychotropic treatment initiated in the month before the breast macrobiopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the reduction in ANXIETY STATE | 1 day
  Evaluation of anxiety before and after RESC session using Spielberger scale

SECONDARY OUTCOMES:
Evaluation of the reduction in ANXIETY STATE | 3 days
  Evaluation of anxiety before and after RESC session using Spielberger scale
Evaluation of the reduction in ANXIETY STATE | 7 days
  Evaluation of anxiety before and after RESC session using Spielberger scale

CONTACTS AND LOCATIONS:
Overall Officials: Celine Lemaire, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No